CLINICAL TRIAL: NCT01844232
Title: A One Year, Open Label, Dose Escalation Study To Evaluate the Long-Term Safety of Arbaclofen Extended Release Tablets (AERT) in Multiple Sclerosis Subjects With Spasticity
Brief Title: One Year, Open Label, Dose Escalation Long-term Safety Study in Multiple Sclerosis (MS) Subjects With Spasticity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: RVL Pharmaceuticals, Inc. (Industry)
Collaborators: Osmotica Pharmaceutical US LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Arbaclofen OS440-3003
Record Dates: First submitted 2013-04-24; First posted 2013-05-01 (Estimated); Last update posted 2022-04-25 (Actual); Status verified 2015-05

CONDITIONS: Multiple Sclerosis; Spasticity
Keywords: Multiple sclerosis; spasticity; arbaclofen
MeSH Terms: conditions — Multiple Sclerosis; Muscle Spasticity | interventions — arbaclofen placarbil

STUDY DESIGN:
Intervention Model Description: All subjects will begin treatment with arbaclofen at 20 milligrams (mg) per day (2 X 10 mg) for two weeks, then increase to 30 mg per day (2 X 15 mg) for two weeks, and then increase to 40 mg per day (2 X 20 mg) based on the Dose Escalation Criteria. Once the subject reaches the Maintenance Dose, they will remain on that dose for approximately 1 year. The Maintenance Dose is the highest tolerated dose, not to exceed 40 mg per day.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arbaclofen Extended Release (ER) Tablets (Experimental): Arbaclofen Extended Release Tablets, 20 mg/day, 30 mg/day or 40 mg/day
  Interventions: Drug: arbaclofen

INTERVENTIONS:
Drug: arbaclofen — Arbaclofen ER tablets, 20 mg, 30 mg and 40 mg
  Other Names: OS440

SUMMARY:
Clinical protocol OS440-3003 is a multicenter, open-label, non-randomized, uncontrolled, dose escalation study to evaluate the safety and tolerability of Arbaclofen Extended Release Tablets over 1 year in Multiple Sclerosis (MS) subjects with spasticity. All subjects in this study will receive arbaclofen in the extended release tablet formulation.

DETAILED DESCRIPTION:
Clinical protocol OS440-3003 is a multicenter, open-label, non-randomized, uncontrolled, dose escalation study to evaluate the safety and tolerability of Arbaclofen Extended Release Tablets (AERT) over 1 year in MS subjects with spasticity. All subjects in this study will receive arbaclofen in the extended release tablet formulation.

All subjects will begin treatment with arbaclofen at 20 milligrams (mg) per day (2 X 10 mg) for two weeks, then increase to 30 mg per day (2 X 15 mg) for two weeks, and then increase to 40 mg per day (2 X 20 mg) based on the Dose Escalation Criteria. Once the subject reaches the Maintenance Dose, they will remain on that dose for approximately 1 year. The Maintenance Dose is the highest tolerated dose, not to exceed 40 mg per day.

In this study, the Up Titration Period begins with Visit 2 and ends when the Maintenance Dose is determined. The Maintenance Period is the time from establishment of the Maintenance Dose until the down-titration visit. For subjects that complete the study, the Maintenance Period is for approximately 1 year in duration. The Down Titration Period will be 2 weeks for subjects on the maintenance dose of 40 mg per day and 1 week for subjects on the maintenance dose of 30 mg per day. There is no down titration phase for subjects on a 20 mg per day maintenance dose.

Subjects for whom the Maintenance Dose is 20 mg per day (i.e., subjects who did not tolerate the 30 mg/ day dose) will begin the 1 year Maintenance Period at Visit 4 and complete the study at Visit 8. Subjects for whom the Maintenance Dose is either 30 mg or 40 mg per day will begin the Maintenance Period at Visit 5 and complete the maintenance portion of the study at Visit 9.

The next portion of the study is down titration. The subjects on the 20 mg per day Maintenance Dose will not have a down-titration. For subjects on the 30 mg per day Maintenance Dose, down-titration will begin at Visit 9 and continue for 1 week. These subjects will return for Visit 10 after the 1 week down-titration. For subjects on the 40 mg per day Maintenance Dose, down titration will begin at Visit 9 and continue for 2 weeks. These subjects will return for Visit 10 after the 2 week down-titration.

Study visits will occur every two weeks until the Maintenance Dose is reached and then study visits will occur every three months with telephone follow-up calls monthly in between visits

ELIGIBILITY:
Inclusion Criteria:

* Patients (male or female) 18 to 70 years of age, inclusive, at the time of the first dose.
* Have an established diagnosis (per McDonald 2005 Criteria, of Multiple Sclerosis Appendix C (either relapsing remitting or secondary progressive course), that manifests spasticity.
* If receiving disease-modifying medications (immunomodulatory treatment), these must have been at a stable dose for at least one (1) months prior to screening, and the subject must be willing to maintain this treatment for the duration of the study.
* If receiving botulinum toxin must be on a stable treatment regimen (e.g. every 12 weeks).
* If receiving phenol or alcohol injections, should have been received 60 days before enrolment in the study.
* Absence of infections and peripheral vascular disease.
* Have a creatinine clearance, as calculated by Glomerular Filtration Rate using the Modification of Diet in Renal Disease (MDRD) formula , greater than 60 milliliters/minute.
* Use of a medically highly effective form of birth control during the study and for 90 days thereafter for women of child-bearing potential (including female subjects and female partners of non-sterile male subjects. .
* Willing to allow his or her general practitioner and consultant, if appropriate, to be notified of participation in the study

Exclusion Criteria:

* Any concomitant disease or disorder that has symptoms of spasticity or that may influence the subject's level of spasticity.
* Inability to rate their level of spasticity or distinguish it from other MS symptoms.
* History of allergy to baclofen.
* Concomitant use of medications that would potentially interfere with the actions of the study medication or outcome variables (Appendix D Prohibited Concomitant Medications)
* Pregnancy, lactation or planned pregnancy during the course of the study and for three months thereafter. (Confirmation that the subject is not pregnant must be established by a negative serum pregnancy test at baseline).
* History of, or current unstable psychiatric disease, or signs and symptoms of significant medical disorders such as severe, progressive, or uncontrolled renal, hepatic, gastrointestinal, hematological, endocrine, immunologic, pulmonary, cardiac or neurological disease which, in the opinion of the investigator, may; put the subject at risk because of participation, influence the result of the study, or affect the subject's ability to participate.
* Seizures requiring medication.
* Current significant cognitive deficit, severe or untreated anxiety, severe or untreated depression.
* Subjects with abnormal micturition that requires indwelling or intermittent catheterization or with lower urinary tract symptoms (LUTS) that result in a score greater than twenty-six (>26) in the Baseline Urinary Symptom Profile© questionnaire.
* Current malignancy or history of malignancy that has not been in remission for more than five years, except effectively treated basal cell skin carcinoma.
* History of substance abuse within the past twelve (12) months.
* Participation in another interventional research study within thirty (30) days of Screening except OS440-3002.
* Patients who are uncooperative or unwilling to sign consent form.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2013-04; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Assessment of Adverse Events | From the beginning of dose titration to end of study (day 393 of dosing)
  Determination of incidence and severity of Adverse Events (AEs), discontinuations due to AEs and discontinuations due to failure of AERT to alleviate spasticity

SECONDARY OUTCOMES:
Determination of Change in Spasticity by Total Number-transformed Modified Ashworth Scale (TNmAS) | From baseline (Day1, Visit 2) to end of treatment (Day 393)
  Change in the total Numeric-transformed Modified Ashworth Scale from baseline to the end of the study (Day 393)

CONTACTS AND LOCATIONS:
Overall Officials: Praveen Tyle, Ph.D., Study Chair — Osmotica Pharmaceutical
Locations (35):
- United States (21):
  - Osmotica Study Site-154, Gilbert, Arizona
  - Osmotica Study Site-158, Phoenix, Arizona
  - Osmotica Study Site-165, Pasadena, California
  - Osmotica Study Site-164, Torrance, California
  - Osomtica Study Site-164, Torrance, California
  - Osmotica Study Site-173, Bradenton, Florida
  - Osmotica Study Site-178, Pompano Beach, Florida
  - Osmotica Study Site-170, Tampa, Florida
  - Osmotica Study Site-179, Northbrook, Illinois
  - Osmotica Study Site-174, Lenexa, Kansas
  - Osmotica Study Site-175, Ann Arbor, Michigan
  - Osmotica Study Site-161, Plainview, New York
  - Osmotica Study Site-151, Charlotte, North Carolina
  - Osmotica Study Site-157, High Point, North Carolina
  - Osmotica Study Site-155, Raleigh, North Carolina
  - Osmotica Study Site-152, Wilmington, North Carolina
  - Osmotica Study Site-156, Dayton, Ohio
  - Osmotica Study Site-163, Philadelphia, Pennsylvania
  - Osmotica Study Site-162, Franklin, Tennessee
  - Osmotica Study Site-171, San Antonio, Texas
  - Osmotica Study Site-166, Vienna, Virginia
- Russia (8):
  - Osmotica Study Site-554, Krasnoyarsk
  - Osmotica Study Site-552, Krasnoyarsk
  - Osmotica Study Site-557, Moscow
  - Osmotica Study Site-556, Moscow
  - Osmotica Study Site-553, Pyatigorsk
  - Osmotica Study Site-551, Saint Petersburg
  - Osmotica Study Site-560, Sestroretsk
  - Osmotica Study Site-555, Tonnel’nyy
- Ukraine (6):
  - Osmotica Study Site-653, Dnipropetrovsk
  - Osmotica Study Site-655, Dnipropetrovsk
  - Osmotica Study Site-651, Donetsk
  - Osmotica Study Site-654, Kharkiv
  - Osmotica Study Site-656, Lviv
  - Osmotica Study Site-657, Poltava